CLINICAL TRIAL: NCT06864819
Title: Role of Phosphatidylethanol in Predicting Perioperative Outcomes of Admitted Patients at UHCMC
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Salim M Hayek, Professor and Vice Chair for Clinical Research, Department of Anesthesiology, University Hospitals Cleveland Medical Center
Other Study IDs: STUDY20240892
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Complications; Alcohol Use Disorder
Keywords: alcohol consumption; surgical outcomes
MeSH Terms: conditions — Postoperative Complications; Alcoholism; Alcohol Drinking | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing elective surgery at UHCMC.: Patients will have a single blood sample sent for PEth testing.
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Patients will have a single blood sample sent for PEth testing, blood draws will happen during standard of care blood draw.

SUMMARY:
This study aims to see if there's a link between a substance called phosphatidylethanol (PEth) and how patients who have surgery at University Hospitals do after surgery. PEth levels reflect the amount of alcohol use by someone over the past few weeks. This study is checking PEth levels on all patients who are planned to stay in the hospital for three or more days after surgery regardless if they drink alcohol. Specifically, it will look at if PEth levels are connected to problems that might come up during and after surgery, like confusion, lung or heart issues, needing blood transfusions, infections, unexpected intensive care unit (ICU) stays, and longer hospital stays. While there are reports of moderate alcohol consumption being good for the heart, there are other data that alcohol consumption can be harmful. Since there's not much information on how drinking alcohol affects health outcomes during and after surgery, especially for patients who are planned to be admitted to the hospital ward or ICU after surgery, this study will hopefully see if PEth levels before surgery can predict how patients do after the surgery.

The inclusion criteria to only include patients who consume alcoholic beverages was an IRB approved modification after already recruiting 1/3 of patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range: 21-79
* 2. Patients undergoing elective surgery at UHCMC with planned ICU admission
* 3. Patients undergoing elective surgery at UHCMC with expected in-hospital admission for three or more days
* 4. Only patients who consume alcoholic beverages on a regular basis.

Exclusion Criteria:

* 1. Patients undergoing same day outpatient surgeries or expected to be admitted less than three days post-operatively
* 2. Subjects who have received a blood transfusion within the past month before surgery
* 3. Pregnant subjects

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery at UHCMC.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Phosphatidylethanol level as measured by blood draw. | Baseline
Length of ICU stay measured in days | Up to 7 days
Length of hospital stay measured in days | Up to 2 weeks
Number of perioperative complications as measured by medical record review. | Up to six months
  Perioperative complications including but not limited to delirium, pulmonary complications, cardiovascular complications, need for transfusion including amount transfused, post-operative infections, unexpected admission to the intensive care unit (ICU) and increased length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Salim Hayek, MD, PhD, Principal Investigator — University Hospitals
Locations (1):
- University Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No